CLINICAL TRIAL: NCT01149382
Title: Humoral Immune Response To Influenza Vaccine In Islet Cell In Transplant Recipients
Brief Title: Immune Response to Influenza Vaccine in Islet Cell Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Assistant Professor, University of Alberta
Other Study IDs: KUOA-03-ITP
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Transplant
Keywords: flu shot; islet cell transplant recipients
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- islet cell transplant recipients

SUMMARY:
Influenza virus is an important cause of morbidity in the transplant population and can lead to viral and bacterial pneumonia. Although the annual influenza vaccine is recommended for organ transplant patients, studies have shown that the standard inactivated influenza vaccine has poor immunogenicity in this population. The investigators plan to test the humoral response to vaccination and look at HLA upregulation

DETAILED DESCRIPTION:
OBJECTIVE AND HYPOTHESIS

* To test the specific humoral response of the influenza vaccine after islet cell transplantation
* To test the production of HLA alloantibodies after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult islet cell transplant recipients
* Able to provide informed consent

Exclusion Criteria:

* Egg allergy
* Previous life-threatening reaction to influenza vaccine (ie Guillain Barre Syndrome)
* Febrile illness in the past two weeks
* Unable to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult islet cell transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
•Seroprotection rate | 3 months
  defined as a post-vaccination titer of ≥1:40

SECONDARY OUTCOMES:
•Seroconversion rate | 3 months
  defined as a 4-fold increase in titer from pre- to post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada